CLINICAL TRIAL: NCT07263919
Title: A Randomized, Controlled, Multi-center Phase II/III Clinical Trial of Perioperative Cadonilimab Combined With Neoadjuvant Chemotherapy in Patients With Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Perioperative Cadonilimab Combined With Neoadjuvant Chemotherapy in Resectable Esophageal Squamous Cell Carcinoma (ESCC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-312
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cadonilimab (dose 1) combined with Cisplatin and Paclitaxel (Experimental)
  Interventions: Drug: Cadonilimab (AK104); Drug: Cisplatin; Drug: Paclitaxel
- Cadonilimab (dose 2) combined with Cisplatin and Paclitaxel (Experimental)
  Interventions: Drug: Cadonilimab (AK104); Drug: Cisplatin; Drug: Paclitaxel
- Cisplatin and Paclitaxel (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cadonilimab (AK104) — Specified doses on specified days.
  Arms: Cadonilimab (dose 1) combined with Cisplatin and Paclitaxel; Cadonilimab (dose 2) combined with Cisplatin and Paclitaxel
Drug: Cisplatin — IV infusion; 75mg/m2
Drug: Paclitaxel — IV infusion; 175mg/m2

SUMMARY:
This is a randomized, controlled, multi-center phase II/III study. All patients are resectable locally advanced thoracic esophageal squamous cell carcinoma (ESCC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of perioperative Cadonilimab combined with neoadjuvant chemotherapy versus neoadjuvant chemotherapy in patients with resectable ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* ≥18 years old and ≤ 75 years (regardless of sex).
* Pathologically confirmed esophageal squamous cell carcinoma, assessed as resectable.
* Adequate pulmonary function.
* Adequate tumor tissue samples.
* ECOG performance status of 0-1.
* Adequate organ function.
* Within 7 days prior to the first dose, women of childbearing potential must have a negative urine or serum pregnancy test and agree to use effective contraception during the study treatment period and for 120 days after the last dose.

Exclusion Criteria:

* Presence of suspected distant metastatic lesions, or locally advanced unresectable disease.
* Histologically confirmed as other pathological types.
* Previous surgery precludes the use of gastric substitution for esophageal reconstruction in the current procedure.
* History of other malignant tumors within the past 5 years.
* Within 4 weeks prior to randomization, presence of conditions such as severe esophagogastric varices, active ulcers, unhealed wounds, gastrointestinal perforation, or intestinal obstruction.
* Active or documented history of inflammatory bowel disease.
* Clinically symptomatic or recurrent pleural, pericardial, or ascitic fluid requiring drainage.
* Uncontrolled concurrent illnesses.
* Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks prior to randomization.
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* History of severe bleeding tendency or coagulation dysfunction.
* Arterial thromboembolic events within 6 months prior to randomization.
* History or current presence of non-infectious pneumonitis/interstitial lung disease requiring systemic glucocorticoids.
* Known psychiatric disorders, drug abuse, or substance addiction.
* Pregnant or lactating women.
* Prior systemic or local antitumor therapy for locally advanced esophageal squamous cell carcinoma.
* Systemic non-specific immunomodulatory therapy within 2 weeks prior to randomization.
* Major surgery or severe trauma within 4 weeks prior to randomization.
* Known allergy to any component of the investigational drug(s).
* Active autoimmune disease requiring systemic treatment within 2 years prior to randomization.
* Active hepatitis B infection.
* Known active tuberculosis.
* Severe infections within 4 weeks prior to randomization.
* History of immunodeficiency or positive HIV test.
* Known active syphilis infection.
* Live vaccination within 4 weeks prior to randomization or planned during the study.
* History of allogeneic organ transplantation or hematopoietic stem cell transplantation.
* Is currently participating in a study of an investigational agent or using an investigational device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) rate as assessed by the investigator | Up to approximately 2 years
  Proportion of subjects with no tumor residue in the primary tumor and regional lymph nodes.
Adverse Event (Phase II stage) | Up to approximately 5 years
  Incidence and severity of adverse events (AEs), rate of delayed surgery, and clinically significant abnormal laboratory findings.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) rate as assessed by the investigator | Up to approximately 2 years
  Proportion of subjects with ≤10% residual live tumor cells as assessed by the investigator.
R0 resection rate | Up to approximately 2 years
  Proportion of subjects with pathologically complete resection of primary tumors
Event Free Survival (EFS) | Up to approximately 5 years
  Time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.
Disease Free Survival (DFS) | Up to approximately 5 years
  Time from surgery to local or distant recurrence, or death due to any cause.
Overall Survival (OS) | Up to approximately 5 years
  Time from randomization until death from any cause.
Overall Response Rate (ORR) | Up to approximately 2 years
  Proportion of subjects with complete response (CR) or partial response (PR) during the neoadjuvant stage.
Disease Control Rate (DCR) | Up to approximately 2 years
  Evaluation of DCR based on RECIST v1.1
Pharmacokinetics (PK) | Up to approximately 2 years
  PK parameters: serum concentrations of Cadonilimab at different point of time
Anti-Drug Antibodies(ADAs) | Up to approximately 2 years
  Proportion of subjects with detectable ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Yan, Principal Investigator — The Second Affiliated Hospital of Air Force Medical University
Locations (1):
- The Second Affiliated Hospital of Air Force Medical University, Xi'an, China